CLINICAL TRIAL: NCT02018289
Title: Effect of Triclosan-coated Suture on Superficial SSI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital General Universitario Elche (Other)
Responsible Party: Principal Investigator, Jaime Ruiz-Tovar, MD, PhD, Professor, Hospital General Universitario Elche
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2013-0010
Record Dates: First submitted 2013-12-17; First posted 2013-12-23 (Estimated); Last update posted 2013-12-23 (Estimated); Status verified 2013-12

CONDITIONS: Surgical Site Infection
Keywords: Triclosan coated suture; Surgical site infection; Fecal peritonitis; Superficial; incisional
MeSH Terms: conditions — Surgical Wound Infection; Surgical Wound

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (2):
- Triclosan (Experimental): Suture of the abdominal wall with triclosan coated suture
  Interventions: Procedure: Triclosan coated suture
- No triclosan (Sham Comparator): Suture of the abdominal wall with the same suture, but without triclosan
  Interventions: Procedure: No triclosan

INTERVENTIONS:
Procedure: Triclosan coated suture — Suture of the abdominal wall with triclosan coated suture
  Arms: Triclosan
Procedure: No triclosan — Suture of the abdominal wall with suture without triclosan coat
  Arms: No triclosan

SUMMARY:
The abdominal closure with triclosan coated suture will reduce superficial surgical site infection.

ELIGIBILITY:
Inclusion Criteria:

* Fecal peritonitis

Exclusion Criteria:

* Perioperative mortality

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2007-10; Primary Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Superficial surgical site infection (SSI) | 60 postoperative days
  SSI will be evaluated in the postoperative course and up to 60 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Ruiz-Tovar, MD, PhD, Principal Investigator — Hospital General Universitario de Elche
Locations (1):
- General University Hospital Elche, Elche, Alicante, Spain